CLINICAL TRIAL: NCT03612050
Title: Development of Meaning Centered Psychotherapy for Palliative Care Patients
Brief Title: Meaning Centered Psychotherapy for Palliative Care Patients (MCP-PC)
Acronym: MCP-PC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fordham University (Other)
Collaborators: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21 NR017728
Record Dates: First submitted 2018-03-15; First posted 2018-08-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Palliative Care
Keywords: Palliative care; Despair; Spiritual well-being

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Placebo Comparator): facilitate any clinical interventions
  Interventions: Behavioral: Meaning Centered Psychotherapy
- Meaning Centered Psychotherapy (Experimental): raise patients' sense of meaning/purpose
  Interventions: Behavioral: Meaning Centered Psychotherapy

INTERVENTIONS:
Behavioral: Meaning Centered Psychotherapy — Manualized, 3-session existential psychotherapy (30-45 minutes/session) with an optional 4th "booster" session. Content focuses on enhancing patients sense of meaning and purpose in life.

SUMMARY:
This randomized, controlled trial evaluates the effectiveness of an adaptation of a well-established brief, structured existential psychotherapy (Meaning Centered Psychotherapy) specifically tailored to the needs of palliative care patients (MCP-PC). Terminally ill patients with cancer who have been hospitalized in a palliative care hospital will be randomly assigned to either MCP-PC or enhanced usual care. Patients will complete a very short battery of self-report measures before the 3-session intervention, and again 2 and 4 weeks later to determine whether treatment has bolstered spiritual and psychological well-being and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Terminal illness with life expectancy of less than 6 months; hospitalized at a palliative care facility in Bronx NY, English speaking

Exclusion Criteria:

* Cognitive impairment or severe psychiatric symptoms that preclude informed consent or participation in treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Spiritual Well Being | Through study completion (approx 6 weeks)
  Overall spiritual well-being as measured through the self-report FACIT Spiritual Well Being scale

SECONDARY OUTCOMES:
Hopelessness | Through study completion (approx 6 weeks)
  Self-report rating scale, the Hopelessness Assessment in Illness scale
Acceptance of Death | Through study completion (approx 6 weeks)
  Subscale derived from the Life Attitude Profile, a self-report measure of meaning and purpose
Health related Quality of life | Through study completion (approx 6 weeks)
  Single item rating of overall quality of life derived from the McGill Quality of Life Questionnaire
Desire for hastened death | Through study completion (approx 6 weeks)
  Abbreviated version of the Schedule of Attitudes towards Hastened Death, a measure of desire for hastened death

CONTACTS AND LOCATIONS:
Overall Officials: Barry Rosenfeld, PhD, Principal Investigator — Fordham University

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request following completion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after completion of data collection.
Access Criteria: Affiliation with medical or university-based research institute

REFERENCES:
- [Background] Rosenfeld B, Saracino R, Tobias K, Masterson M, Pessin H, Applebaum A, Brescia R, Breitbart W. Adapting Meaning-Centered Psychotherapy for the palliative care setting: Results of a pilot study. Palliat Med. 2017 Feb;31(2):140-146. doi: 10.1177/0269216316651570. Epub 2016 Jul 21. PMID 27435603